CLINICAL TRIAL: NCT04522245
Title: Evaluation of Brain Activity Changes After a Behavior Change Weight Loss Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noom Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Andreas Michaelides, Chief of Psychology, Noom Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00042660
Record Dates: First submitted 2020-08-04; First posted 2020-08-21 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Obesity; Behavior, Health; Weight Loss
Keywords: EEG, mhealth, weight loss, CBT, cognitive behavior therapy
MeSH Terms: conditions — Obesity; Health Behavior; Weight Loss; Color Vision Defects | interventions — Case-Control Studies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Matched control group (Noom-branded 'healthy eating' short guide on weight loss).
  Interventions: Other: Matched Control
- Noom Health Weight Program (Experimental)
  Interventions: Behavioral: Noom Healthy Weight; mobile behavior change program for weight loss.

INTERVENTIONS:
Behavioral: Noom Healthy Weight; mobile behavior change program for weight loss. — The mobile cognitive behavior change program follows guidelines from the Obesity Society's "2013 Guidelines for the Management of Overweight and Obesity in Adults" NIH "Practical Guide on the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults".
  There are 52 weeks of curriculum with 1-3 articles to read per day. Users are requested to perform weight logging once daily and food logging after each meal. Users are assigned human coaches and are able to interact with them via in-app messaging or phone communication. Users are also assigned to support groups via in-app messaging.
  Arms: Noom Health Weight Program
Other: Matched Control — Matched control group (Noom-branded 'healthy eating' short guide on weight loss).
  Arms: Control

SUMMARY:
The aim of this study is to compare brain changes in individuals with overweight or obesity enrolled in either the Noom Healthy Weight program or a matched control. The study objectives (primary and secondary) are to measure brain change reported as ERP and EEG data over a 16-week timeframe. Additionally, we will explore changes in the default mode network (resting-state asymmetry in EEG measurements), changes in executive functioning, quality of life, mood, and salivary markers as they relate to EEG data.

ELIGIBILITY:
Inclusion criteria:

* Each subject must be able to understand and provide informed consent
* Between the ages 18-60 years
* Self-report of good health
* Overweight or obesity (BMI ≥ 25)
* Able to meet our criteria of adherence to the program
* Able to attend in-person visit in Long Island, NY

Exclusion criteria:

* Inability or unwillingness to give written informed consent or comply with the study
* Visual impairment that cannot be corrected with glasses or contact lenses
* Any indication of drug, alcohol or medicine abuse.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
* Presence of a brain injury, psychiatric disorders, seizure disorders, and other neurological conditions
* Reported eating disorder
* Currently pregnant or 6 months postpartum
* Planning to become pregnant within the next 5 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Change in Flanker task performance: Intervention vs control | 16 weeks
  Change in amplitude and latency in conflict monitoring stage at 16 weeks
Change in behavioral inhibition | 16 weeks
  Change from baseline Flanker task performance at 16 weeks
Change in behavioral inhibition | 16 weeks
  Change from baseline n-back task performance at 16 weeks
Change in behavioral inhibition | 16 weeks
  Change from baseline Stroop test at 16 weeks

SECONDARY OUTCOMES:
Change in EEG data: Successful intervention (5% weight loss) in higher engagement subgroup (successful program completers) vs control | 16-week
  Task-specific event-related potential (ERP) peak amplitude and latency for channels and
  * Task-specific event-related potential (ERP) peak amplitude and latency for channels and cortical ROIs
  * Event-related spectral perturbation (time x frequency power) for channels and cortical ROIs
  * Mean and relative power spectral density measures for each frequency band + select ratios, for channels and cortical ROIs
  * Brain connectivity between cortical ROIs
Comparison of EEG data in program starters to successful program completers | 16-week
  * Task-specific event-related potential (ERP) peak amplitude and latency for channels and cortical ROIs
  * Event-related spectral perturbation (time x frequency power) for channels and cortical ROIs
  * Mean and relative power spectral density measures for each frequency band + select ratios, for channels and cortical ROIs
  * Brain connectivity between cortical ROIs
Within-subject comparison for EEG data | 16-week
  * Task-specific event-related potential (ERP) peak amplitude and latency for channels and cortical ROIs
  * Event-related spectral perturbation (time x frequency power) for channels and cortical ROIs
  * Mean and relative power spectral density measures for each frequency band + select ratios, for channels and cortical ROIs
  * Brain connectivity between cortical ROIs

OTHER OUTCOMES:
Change in Positive and Negative Affect Schedule (PANAS-SF) | 16-week
  Explore measure as it relates to change in EEG data
Change in quality of life outcome measure scoring (PROMIS-29) | 16-week
  Explore measure as it relates to change in EEG data
Change in eating behavior measure scoring (Three-Factor Eating Questionnaire) | 16-week
  Explore measure as it relates to change in EEG data
Change from baseline salivary stress marker at 16 weeks | 16-week
  Cortisol
Change from baseline salivary tumor necrosis factor alpha at 16 weeks | 16-week
  TNF-a
Change from baseline salivary interleukin-6 at 16 weeks | 16-week
  IL-6
Change from baseline blood pressure (systolic/diastolic) at 16 weeks | 16-week

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michaelides, PhD, Principal Investigator — Chief of Psychology
Locations (1):
- Focus Feedback, Commack, New York, United States

IPD SHARING:
Plan to Share IPD: No